CLINICAL TRIAL: NCT00596401
Title: The Effect of Helicobacter Pylori Eradication on the Development of Gastric Cancer and the Medical Care Cost in Iijima Town
Brief Title: The Preventive Effect of Helicobacter Pylori Eradication on the Development of Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Digestive Disease Center, Showa Inan General Hospital
Other Study IDs: sihp20076
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Helicobacter Pylori; Eradication; Gastric Cancer; Medical Care Cost
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: HP eradication group
- 2: No eradication group
- 3: No Hp group

SUMMARY:
Recently, the preventive effect of Helicobacter pylori (Hp) eradication treatment on the incidence of gastric cancer has been reported. By Hp eradication treatment being performed for Hp-infected people in Iijima town, we will evaluate whether the incidence of gastric cancer and/or the medical care cost can be reduced as compared with those in the previous years.

ELIGIBILITY:
Inclusion Criteria:

* People who live in Iijima town at their age of 19 to 69 years

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who live in Iijima town
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
the annual incidence of gastric cancer in Iijima town | 10 years

SECONDARY OUTCOMES:
The annual medical care cost in Iijima town | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Akira Horiuchi, M.D., Study Director — Showa Inan General Hospital
Locations (1):
- Showa Inan General hospital, Komagane, Nagano, Japan